CLINICAL TRIAL: NCT04453748
Title: The Assessment of the Prevalence, Clinical Course and Treatment of COVID-19 Complications
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Silesian Centre for Heart Diseases (Other)
Collaborators: Medical Research Agency, Poland (Other Government); Medical University of Silesia (Other)
Responsible Party: Principal Investigator, Mariusz Gasior, Prof., Silesian Centre for Heart Diseases
Other Study IDs: COVID-19 Complications Study
Record Dates: First submitted 2020-05-21; First posted 2020-07-01 (Actual); Last update posted 2020-09-30 (Actual); Status verified 2020-09

CONDITIONS: COVID-19; Coronavirus Infection; Sars-CoV2; Complications
Keywords: COVID-19; Sars-CoV2; Complications
MeSH Terms: conditions — COVID-19; Coronavirus Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Biospecimen Retention: Samples Without DNA — Blood, urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- COVID-19 convalescents: People who recovered from COVID-19: have no symptoms and no SARS-Cov2 RNA in PCR
  Interventions: Other: Complex diagnostic panel

INTERVENTIONS:
Other: Complex diagnostic panel — Complex, multidisciplinary diagnostic panel, including blood, imaging and functional tests.

SUMMARY:
SAR-Cov-2 infection and its clinical manifestation known as COVID-19 beside the respiratory and lung involvement may include the cardiovascular system, the nervous system and the liver. In the acute phase of the disease, all of these conditions may be life-threatened. As a result, after the acute phase of COVID-19, early complications may be observed, including heart, lungs, brain, muscles and liver. A few papers to date have been reported of myocarditis, ventricular arrhythmias, post-inflammatory changes in the lung and liver, as well as ischemic changes in the brain, diseases of skeletal muscle, which may have adverse prognostic effects. Due to the extent of the pandemic, the severity of the complications and the expected high complications' prevalence in the early post-recovery period, a study was designed to determine the extent of the problem of early complications after COVID-19. Complex cardiological, pulmonary, neurological and hepatological diagnostics are planned, including laboratory, imaging and functional tests. The results obtained, in addition to determining the scale of the problem, will allow the selection of studies that optimally identify patients with early complications. The purpose of this procedure is to enable rapid treatment of diseases that are complications of SARS-COV-2 infection. An additional aspect raised in the project will be the issue of psychiatric disorders (anxiety, depression, post traumatic disorders).

The main three purposes of the study include:

1. the assessment of prevalence of particular complications after COVID-19.
2. identification of the demographic and clinical risk factors of COVID-19 complications
3. determining the diagnostic tests which are sufficient to detect early complications of COVID-19

ELIGIBILITY:
Inclusion Criteria:

1. SARS-Cov-2 RNA confirmed by the PCR method in the acute phase of disease.
2. Presence of the clinical symptoms associated with COVID-19 in the acute phase of disease
3. Two negative results of SARS-COV-2 PCR test following the 7-day period of quarantine
4. Informed consent

Exclusion Criteria:

1. Any symptoms of infection during the quarantine
2. Lack of patient's consent
3. Lack of possibility of travelling to the hospital for tests

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who recovered from COVID-19 in Silesia, Poland.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-06-08 (Actual); Primary Completion 2021-10-31 (Estimated); Study Completion 2021-11-30 (Estimated)

PRIMARY OUTCOMES:
Prevalence of COVID-19 complications | 2 months
  Complications include pulmonary, cardio-vascular, neurological, hepatologic and psychiatric disordes that might be linked to the COVID-19.
  The diagnostic tests: blood tests, transthoracic echocardiography, spirometry, high-resolution computed tomography, neurological examination, liver ultrasonography and elastography, vasular ultrasonography (veins and arteries), psychiatric questionnairies

SECONDARY OUTCOMES:
Assessment of risk factors of COVID-19 complications | 2 months
  Analysis which demographic and clinical parametrs were associated with particular COVID-19 complication.
  Statistical analysis of relation between clinical parameters before and during COVID19 and the occurence of COVID19 complications

CONTACTS AND LOCATIONS:
Locations (1):
- Silesian Centre for Heart Disease, Zabrze, Silesian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Pudlo R, Jaworska I, Szczegielniak A, Niedziela J, Kulaczkowska Z, Nowowiejska-Wiewiora A, Jaroszewicz J, Gasior M. Prevalence of Insomnia in the Early Post-COVID-19 Recovery Period. Int J Environ Res Public Health. 2022 Oct 31;19(21):14224. doi: 10.3390/ijerph192114224. PMID 36361102